CLINICAL TRIAL: NCT07214428
Title: Effects of Grape Powder on Psychological Distress and Gut Microbiota in College Students (FTGP2025)
Brief Title: Effects of Grape Powder on Psychological Distress and Gut Microbiota in College Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: California Table Grape Commission (Other)
Responsible Party: Principal Investigator, Guojun Wu, Ph.D., Assistant Research Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro2025001394
Record Dates: First submitted 2025-10-01; First posted 2025-10-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gut Microbiota; Psychological Distress
Keywords: Table grape; Gut Microbiota; psychological distress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- freeze-dried table grape powder (FTGP) (Experimental): Drink a daily supplement containing FTGP for 4 weeks
  Interventions: Dietary Supplement: freeze-dried table grape powder
- Placebo (Placebo Comparator): Drink a daily supplement containing a placebo for 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: freeze-dried table grape powder — 48g freeze-dried table grape powder/day for 4 weeks
  Arms: freeze-dried table grape powder (FTGP)
Dietary Supplement: Placebo — 48g placebo/day for 4 weeks
  Arms: Placebo

SUMMARY:
The goal of this trial is to investigate the effect of freeze-dried table grape powder (FTGP) on psychological distress and gut microbiota in college students. The main questions it aims to answer are:

Does FTGP reduce anxiety, depression, and perceived stress? Does FTGP improve the gut microbiota? Researchers will compare FTGP to a placebo to see how FTGP affects psychological distress and gut microbiota.

Participants will:

Drink a daily supplement containing FTGP or a placebo for 4 weeks. Record consumption of grape powder or placebo in a compliance log. Complete surveys and provide stool samples. Three in-person visits.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years old
* Able to give written informed consent.
* BMI 18.5-24.9 kg/m2
* Healthy (self-reported)
* Can read and speak English

Exclusion Criteria:

* Currently taking medications that interfere with polyphenol
* Currently using or have used antibiotics continuously for >3 days within 3 months prior to enrollment
* Have had surgery involving the intestinal lumen within the last 30 days
* Have a documented diagnosis of celiac disease or/and inflammatory bowel diseases
* Are pregnant or breastfeeding
* Have prediabetes and diabetes
* Have had bariatric surgery
* Are immunocompromised ( e.g., cancer treatment, bone marrow/organ transplant, immune deficiency, or poorly controlled HIV/AIDS)
* Are unable to provide consent
* Are hospitalized,
* Have a history of or current alcohol, drug, or medication abuse (self-reported),
* Have contraindication to any substance in the investigational product or who are currently enrolled in other interventional trials

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Scale -14 | baseline (1st), week 4 (2nd) and week 5 (3rd)
  HAMA-14 is one of the earliest and most widely used clinical scales for measuring the severity of a patient's anxiety. It has 14 items, each reflecting a cluster of anxiety symptoms. Total range: 0 to 56, with higher scores indicating greater severity of anxiety
17-item of Hamilton Depression Rating Scale | baseline (1st), week 4 (2nd) and week5 (3rd)
  HAMD-17 is one of the most widely used clinician-administered scales for measuring the severity of a patient's depression. It has 17 items, each covering symptoms of depression across mood, physical, and cognitive domains. With higher scores indicating greater severity of depression.
10-item of Perceived Stress Scale | baseline (1st), week 4 (2nd) and week5 (3rd)
  PSS-10 is one of the most widely used psychological instruments for measuring the perception of stress. It has 10 items, each reflecting how unpredictable, uncontrollable, and overloaded respondents find their lives during the past month. Total range: 0 to 40, with higher scores indicating greater perceived stress.

SECONDARY OUTCOMES:
Shannon Index of gut microbiota | baseline (1st), week 4 (2nd) and week5 (3rd)
  Changes in gut microbiota will be assessed from stool samples using 16S rRNA gene sequencing. Alpha diversity will be calculated using Shannon Index. This measure will characterize whether the intervention alters gut microbial diversity in each subject.
Beta diversity of gut microbiota | baseline (1st), week 4 (2nd) and week 5 (3rd)
  Changes in gut microbiota will be assessed from stool samples using 16S rRNA gene sequencing. Beta diversity will be calculated using Bray Curtis distance between samples. This measure will characterize whether and how the intervention alters gut microbial communities.
fecal short chain fatty acid | baseline (1st), week 4 (2nd) and week5 (3rd)
  fecal short chain fatty acid will be measured by GC-MS

CONTACTS AND LOCATIONS:
Overall Officials: Guojun Wu, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Department of Biochemistry and Microbiology, School of Environmental and Biological Sciences, Rutgers, The State University of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
IPD might not be shared according to the consent form.

DOCUMENTS (1):
  • Informed Consent Form (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT07214428/ICF_000.pdf